CLINICAL TRIAL: NCT02027077
Title: A Randomized Controlled Trial Evaluating a Small Change Approach to Preventing Long Term Weight Gain in Overweight and Obese Adults
Brief Title: Evaluating a Small Change Approach to Preventing Long Term Weight Gain in Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Bob Ross, Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ross2013
Record Dates: First submitted 2014-01-02; First posted 2014-01-03 (Estimated); Last update posted 2019-01-18 (Actual); Status verified 2017-04

CONDITIONS: Obesity; Prevention of Weight Gain
Keywords: physical activity; diet; small change; behavior change
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Control group
  Interventions: Behavioral: Control group
- Lifestyle counseling (Active Comparator): Behavioral intervention group
  Interventions: Behavioral: Lifestyle counselling

INTERVENTIONS:
Behavioral: Control group — No prescribed intervention/ Participants asked to follow normal initiatives to engage in physical activity a healthful diet behaviors for the duration of the intervention
  Arms: Control group
Behavioral: Lifestyle counselling — Participants will follow a prescribed behavioral intervention program seeking small changes in both physical activity and diet for the duration of the intervention.
  Arms: Lifestyle counseling

SUMMARY:
Obesity is a major risk factor for disease and a public health problem. Recent information suggests that while it is possible for most overweight adults to lose a substantial amount of weight, maintaining the weight loss for any extended time (2 to 3 years) is very difficult. This is because trying to maintain big changes in exercise and/or eating behaviour is very difficult in today's environment that makes sustain big changes in behaviour (Example: eat allot less or exercise allot more) very hard. In fact at this time health professionals are unsure of how best to help overweight adults maintain big behavioral changes for long periods of time. In response, we propose that making smaller changes in eating and exercise habits every day may be possible in today's environment and if so, small weight changes may be possible to maintain for long periods of time. This study is designed to assess whether making small changes in eating and exercise behavior will be associated with sustained weight loss over three (3) years. The results of the study may have important implications for development of public health messages and clinical guidelines for prevention and treatment of obesity through small changes in both exercise and eating habits.

DETAILED DESCRIPTION:
The prevalence of obesity and associated morbidity among Canadian adults is already high and increasing. Prevalence estimates for overweight determined from measured height and weight now exceeds 62 % in Canadian adults1; approximately 15.5 million Canadian adults are now overweight and obese1. Obesity is associated with a wide range of health outcomes from co-morbidities including type 2 diabetes, cardiovascular disease and certain cancers, to psychiatric disorders such as depression1. Direct costs attributed to obesity in Canada range from 4.6 to 7.1 billion dollars annually1. Despite agreement concerning the urgent need to address the obesity problem; few strategies have been successful on a wide scale basis. Past efforts to achieve and sustain weight loss have not been particularly successful. We3 and others4 have repeatedly demonstrated in randomized controlled trials that most adults are not able to sustain the major changes in behaviour that are required to maintain weight loss long term. Thus, although it is an admirable goal to substantially reduce the number of overweight or obese Canadians, this goal may be totally out of reach in the short term. The question then is what can be done to address the obesity problem now? We propose that a reasonable start point in addressing the obesity problem is to develop behavioural goals for prevention of weight gain. This strategy can at least keep the problem from getting worse and at best, can reduce obesity rates over time.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 25 and 65 years of age.
* Overweight or Class I or Class II BMI.
* Walk without assistance.
* Commit to a schedule of assessment visits

Exclusion Criteria:

* Physical impairment which would make the intervention very difficult, or unsafe according to the patient's physician including history of myocardial infarction, stroke, coronary bypass surgery or angioplasty in the last 6 months; peripheral artery disease, unstable angina or ischemia.
* Enrolled within past year in a formal weight loss program
* Reported losing greater than 5% of current body weight in the previous 6 months,
* Smoking
* Plans to move from the area,
* Participating in another research study.
* Clinically judged to be unsuitable for participation or adherence as determined by the participants physician
* Inability or unwillingness to provide informed consent.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2014-02; Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | 2 years

SECONDARY OUTCOMES:
Waist Circumference | 2 years
Physical Activity | 2 years
  Measured by pedometer and self-report
Total and regional body composition measures | 2-years
  Total fat, abdominal subcutaneous and visceral fat and total lean mass measured by DXA.

OTHER OUTCOMES:
Cardiometabolic risk factors | 2 years
  Insulin, glucose, systolic and diastolic blood pressure, triglycerides, LDL- and HDL-cholesterol) , LDL-cholesterol and Apolipoprotien A1, B and inflammatory markers and adipokines including C-reactive protein, IL-6, TNF-alpha and adiponectin.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ross, PhD, Principal Investigator — Queen's University
Locations (1):
- School of Kinesiology and Helath Studies, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Ross R, Latimer-Cheung AE, Day AG, Brennan AM, Hill JO. A small change approach to prevent long-term weight gain in adults with overweight and obesity: a randomized controlled trial. CMAJ. 2022 Mar 7;194(9):E324-E331. doi: 10.1503/cmaj.211041. PMID 35256388